CLINICAL TRIAL: NCT07144020
Title: Donor Derived CD117 CAR-T Cells in the Treatment of Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Donor Derived CD117 CAR-T Cells in the Treatment of R/R Acute Myeloid Leukemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Yake Biotechnology Ltd. (Industry)
Responsible Party: Principal Investigator, He Huang, Principal Investigator, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TXB2024010
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: CD117 CAR-T
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cells（ chimeric antigen receptor T cells） (Experimental): Dose escalation follows the standard 3+3 dose escalation design. A total of 3 dose levels are set for subjects.
  Interventions: Biological: CD117 CAR T-cells

INTERVENTIONS:
Biological: CD117 CAR T-cells — Each subject receive CD117 CAR T-cells by intravenous infusion
  Other Names: CD117 CAR T-cells injection

SUMMARY:
A Clinical Study on the Safety and Effectiveness of Donor Derived CD117 CAR-T Cell in the treatment of Relapsed/Refractory Acute Myeloid Leukemia

DETAILED DESCRIPTION:
This is a single-arm, open-label, dose-escalation clinical trial to evaluate the safety and efficacy of CD117 CAR-T Cell in patients with relapsed or refractory acute myeloid leukemia. It is planned to enroll 15-50 participants in this trial.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with a histologically or immunophenotypically confirmed diagnosis of CD117-positive Acute Myeloid Leukemia (AML).
* 2. Diagnosis must meet the 2016 WHO classification criteria for AML and fulfill the definitions for relapsed or refractory disease per the *Chinese Guidelines for the Diagnosis and Management of Relapsed/Refractory Acute Myeloid Leukemia (2017 Edition)*, with no available suitable standard therapeutic options or registered clinical trials.
* a). Relapsed AML: Defined as the reappearance of leukemic blasts in the peripheral blood, bone marrow blast count >5% (when assessed morphologically, after excluding regenerative changes post-consolidation chemotherapy), or development of extramedullary disease after achieving a Complete Remission (CR).
* b). Refractory AML (meeting at least one criterion): Failure to achieve CR following two cycles of standard induction therapy in newly diagnosed patients; relapse within 12 months after CR following consolidation therapy; relapse beyond 12 months that fails to respond to conventional salvage chemotherapy; ≥2 relapses; or persistent extramedullary leukemia.
* 3. Presence of >5% bone marrow blasts (by morphology) and/or >1% (by flow cytometric analysis).
* 4. Total bilirubin ≤1.5 × ULN (≤51 μmol/L) ALT and AST ≤3 × ULN Serum creatinine ≤1.5 × ULN (≤176.8 μmol/L)
* 5. Left ventricular ejection fraction (LVEF) ≥50% as assessed by echocardiography.
* 6. Oxygen saturation ≥92% on room air.
* 7. Life expectancy ≥3 months.
* 8. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
* 9. For patients of childbearing potential: Agreement to use highly effective contraception from screening, throughout the study treatment period, and for at least 6 months after the cell infusion (due to unknown risks to the fetus).
* 10. Voluntary participation, understanding of the study procedures, and provision of written informed consent by the patient or their legally authorized representative.

Exclusion Criteria:

* 1. Patients with the history of epilepsy or other CNS disease;
* 2. Patients with prolonged QT interval time or severe heart disease;
* 3. Active infection with no cure;
* 4. Active infection of hepatitis B virus or C virus ;
* 5. Before using any gene therapy products;
* 6. The proiferation rate is less than 5 times response to CD3/CD28 co-stimulation signal;
* 7. Suffering from other uncontrolled diseases that the researchers consider unsuitable for joining;
* 8. Infected with AIDS virus;
* 9. Any situation that researchers believe may increase the risk to the subjects or interfere with the trial results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-05 (Estimated); Primary Completion 2028-09-05 (Estimated); Study Completion 2028-09-05 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | Up to 28 days after Treatment
  Adverse events assessed according to NCI-CTCAE v5.0 criteria
Incidence of treatment-emergent adverse events (TEAEs) | Up to 2 years after Treatment
  Incidence of treatment-emergent adverse events [Safety and Tolerability]

SECONDARY OUTCOMES:
Complete response (CR), and complete response with incomplete hematologic recovery (CRi) | Up to 12 weeks after CAR-T infusion
  The proportion of patients with CR (complete response) /CRi (complete response with incomplete blood cell recovery) and PR (partial response).
Duration of remission ,DOR | Up to 1 years after CAR-T infusion
  The time from CR/CRi and PR to disease relapsed or death due to disease progression after CAR-T infusion
Overall survival, OS | Up to 1 years after CAR-T infusion
  The time from CAR-T infusion to death due to any cause
Leukemia-Free Survival, LFS | Up to 2 years after Treatment
  The time from CAR-T infusion torecurrence or metastasis

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The first affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No